CLINICAL TRIAL: NCT03337438
Title: Alcohol and Health: Personalized Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Principal Investigator, Emma Brett, Graduate Student, Oklahoma State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AS1770
Record Dates: First submitted 2017-10-27; First posted 2017-11-09 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Alcohol Drinking; Alcohol Consumption, Youth
MeSH Terms: conditions — Alcohol Drinking; Underage Drinking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Values-PFI (Other)
  Interventions: Other: Personalized Feedback Intervention with Values
- Traditional-PFI with values assessment (Other)
  Interventions: Other: Personalized Feedback Intervention Traditional
- Traditional PFI no values assessment (Other)
  Interventions: Other: Personalized Feedback Intervention Traditional

INTERVENTIONS:
Other: Personalized Feedback Intervention with Values — The PFI with values will include information commonly included in personalized feedback interventions for alcohol use, such as norms information and drinking profile, as well as feedback on three of the assessed values that are highly important to the participant.
  Arms: Values-PFI
Other: Personalized Feedback Intervention Traditional — This PFI will include information on drinking profile, norms, behavioral strategies used while drinking, and practical costs related to drinking reframed as monetary values and caloric values.
  Arms: Traditional PFI no values assessment; Traditional-PFI with values assessment

SUMMARY:
Heavy episodic drinking (HED) among college students remains a concern within the U.S., as rates of HED are still high in this population. Though a variety of brief motivational interventions for alcohol use in college students have demonstrated significant effects, these effects are often small and not consistently maintained over time. Personalized feedback interventions (PFIs) are a particularly promising approach, as these are often acceptable to college students, as well as low-cost, and easy to disseminate. Though presentation of interperson discrepancy via descriptive and injunctive norms has shown consistent effects within PFIs and received much attention in the literature, intraperson, or ideal-actual self discrepancies, has largely been ignored. Drawing from cognitive dissonance theory, self-regulation theory, and motivational interviewing, the current study aims to evaluate the efficacy of an alcohol PFI with a values component to incorporate ideal-self discrepancy into a typical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must be able to speak and read English
* Must report consuming alcohol in a typical week over the past month

Exclusion Criteria:

* Must not deny drinking within the past month
* Non-English speaking
* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-10-22 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | one-month post baseline
  measured by drinks per week
Alcohol consequences | one month post-baseline
  measured by the BYAACQ to determine number of consequences experienced in the past month post-baseline
Value-behavior discrepancy for values related to alcohol use | one month post-baseline
  Measured by the VLQ-A to measure change in behavioral consistency with values specifically related to alcohol use one month post-baseline

SECONDARY OUTCOMES:
Perceptions of norms | one month post-baseline
  Perceptions of descriptive norms will be more accurate one month post-baseline
Trait mindfulness | one month post-baseline
  Levels of mindfulness as measured by the FFMQ will be measured at both time points

CONTACTS AND LOCATIONS:
Locations (1):
- North Murray Hall Oklahoma State University, Stillwater, Oklahoma, United States